CLINICAL TRIAL: NCT06403228
Title: The Effect of Mindfulness Based Structured Nursing Interventions on Mental Health Parameters of High Risk Pregnant Women
Brief Title: The Effect of Mindfulness Based Structured Nursing Interventions on Mental Health Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Elcin Alacam, MSc, Nurse, Principal Investigator, Mersin Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MersinUniversityNursingFaculty
Record Dates: First submitted 2024-05-02; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Mindfulness; Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The intervention group participated in a mindfulness-based structured nursing interventions program planned for a total of eight days, 60 minutes each day, led by Elçin Alaçam, who has a Mindfulness Institute-approved certificate. The mindfulness-based structured nursing interventions program was structured for 8 days, taking into account the literature and the characteristics of high-risk pregnant women such as length of hospitalization.
  Interventions: Other: Mindfulness Based Structured Nursing Interventions
- Control Group (No Intervention): No intervention was applied to the control group. Data were collected from the control group simultaneously with the study group.

INTERVENTIONS:
Other: Mindfulness Based Structured Nursing Interventions — In the study, 8 days of mindfulness-based structured nursing interventions were applied to high-risk pregnant women. The program lasts 60 minutes each day. The program includes short body scanning meditation, breath awareness meditation, sitting meditation, compassion meditation.
  Arms: Experimental Group

SUMMARY:
This randomized controlled study evaluate the effect of mindfulness-based structured nursing interventions on the mental health parameters of risky pregnant women. The hypothesis of this study is that mindfulness-based structured nursing interventions has an effect of the state-trait anxiety, perceived stress, depression on high risk pregnant women.

DETAILED DESCRIPTION:
Methods: This study, was carried out in three phases. In the first phase, the views and experiences of high-risk pregnant women about being treated in the hospital and in the third phase, their views and experiences about the intervention were determined through individual in-depth interviews.In the second phase, 40 high risk pregnant women were randomly assigned to the study and control groups. The study group (n = 19) received 8 days of mindfulness-based structured nursing interventions. The control group (n = 21) did not receive any intervention. Results were collected through data collection forms before the mindfulness-based structured nursing interventions, after the mindfulness-based structured nursing interventions is completed.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65
* Able to read and understand Turkish
* Written informed consent was obtained before participation in the study
* Diagnosed with a risky pregnancy and treated in hospital
* Not receiving any other psychological therapy
* No prior meditation experience
* The participants do not have any physical/mental disability or limitation and disease that would prevent them from participating in the program

Exclusion Criteria:

* Under 18 years old
* Cant read and understand Turkish
* Pregnant women who have not been diagnosed a risky pregnancy or treated in hospital
* Meditation or psychological therapy experiences before the study
* The participants who left the program voluntarily or participating in less than 70% of the eight-day program

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — High risk pregnant women
Enrollment: 40 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Anxiety was assessed using the State-Trait Anxiety Scale | Change from before intervention up to after intervention, on average 1 week upon completion of the intervention.
  The total score obtained from both scales varies between 20 and 80. It states that 0-19 points mean no anxiety, 20-39 points mean mild, 40-59 points mean moderate, 60-79 points mean severe anxiety, and individuals with a score of 60 and above need professional help.
Stress was assessed using the Perceived Stress Scale | Change from before intervention up to after intervention, on average 1 week upon completion of the intervention.
  Total scores range from 0 to 40, with higher scores indicating higher perceived stress. Scores ranging from 0-13 would be considered low stress, from 14-26 moderate stress, and from 27-40 high perceived stress.
Depression was assessed using the Edinburgh Postnatal Despression Scale | Change from before intervention up to after intervention, on average 1 week upon completion of the intervention.
  Each item is scored 0-3 with a maximum total score of 30. Higher scores indicate a greater severity of symptoms. The most commonly-used cut-offs are ≥ 10 to indicate minor depression and ≥ 13 to indicate major depression.

SECONDARY OUTCOMES:
Semi-structured Individual In-Depth Interview Questionnaire I | Before the intervention, on average 1 week upon completion of the intervention.
  Semi-structured Individual In-Depth Interview Questionnaire I was created by the researcher in order to evaulate the views and experiences of high risk pregnant women regarding hsopitalization.
Semi-structured Individual In-Depth Interview Questionnaire II | After the intervention, on average 1 week upon completion of the intervention.
  Semi-structured Individual In-Depth Interview Questionnaire II was created by the researcher in order to evaulate the views and experiences of high risk pregnant women in the study group regarding intervention program.

CONTACTS AND LOCATIONS:
Overall Officials: Mualla Yılmaz, Professor, Study Director — Mersin University
Locations (1):
- Mersin University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No